CLINICAL TRIAL: NCT00613314
Title: Clinical EvaluatioN of TElmisartan-based Antihypertensive Regimen (CENTER)
Brief Title: Clinical EvaluatioN of TElmisartan-based Antihypertensive Regimen
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Other Study IDs: 502.532
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Results first posted 2010-03-05 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-04

CONDITIONS: Hypertension; Metabolic Syndrome X
MeSH Terms: conditions — Hypertension; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
To determine the efficacy and safety of telmisartan-based treatment among patients with metabolic syndrome in actual setting in Philippines.

ELIGIBILITY:
Inclusion Criteria:

* Age > 45 years
* Increased waist circumference (>88.9cm [>35in] men, >78.7cm [>31in] for women)
* Elevated triglycerides (>150mg/dl)
* Low HDL cholesterol (<40mg/dl in men, <50mg/dl in women)
* Hypertension (>130/>85mmHG)
* Impaired fasting glucose (>110mg/dl) (8)
* Hypertensive patient assessed to benefit from telmisartan based treatment

Exclusion Criteria:

* Hypersensitivity to telmisartan, hydrochlorothiazide (HCTZ) and its excipients
* <3 months myocardial infarction (MI), stroke or severe heart failure

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 15268 (Actual)
Dates: Start 2007-06; Primary Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (122):
- Philippines (122):
  - Boehringer Ingelheim Investigational Site, Alaminos City, Pangasinan
  - Boehringer Ingelheim Investigational Site, Angeles City
  - Boehringer Ingelheim Investigational Site, Angeles City, Pampanga
  - Boehringer Ingelheim Investigational Site, Antipolo City, Rizal
  - Boehringer Ingelheim Investigational Site, Atabay, San Jose
  - Boehringer Ingelheim Investigational Site, Bacoor, Cavite
  - Boehringer Ingelheim Investigational Site, Baguio City, Benguet
  - Boehringer Ingelheim Investigational Site, Balanga City, Bataan
  - Boehringer Ingelheim Investigational Site, Baliuag, Balacan
  - Boehringer Ingelheim Investigational Site, Baliuag, Bulacan
  - Boehringer Ingelheim Investigational Site, Bangued, Abra
  - Boehringer Ingelheim Investigational Site, Batac, Ilocos Norte
  - Boehringer Ingelheim Investigational Site, Batangas City, Batangas
  - Boehringer Ingelheim Investigational Site, Batangas City. Batangas
  - Boehringer Ingelheim Investigational Site, Bauan Batangas
  - Boehringer Ingelheim Investigational Site, Bautista, Pangasinan
  - Boehringer Ingelheim Investigational Site, Binan, Laguna
  - Boehringer Ingelheim Investigational Site, Bocaue, Bulacan
  - Boehringer Ingelheim Investigational Site, Butuan
  - Boehringer Ingelheim Investigational Site, Butuan City, Agusan Del Norte
  - Boehringer Ingelheim Investigational Site, Cabanatuan City, Nueva Ecija
  - Boehringer Ingelheim Investigational Site, Cagayan de Oro City, Misamis Oriental
  - Boehringer Ingelheim Investigational Site, Cagayan de Oro City, Misamis
  - Boehringer Ingelheim Investigational Site, Cagayan de Oro, Misamis Oriental
  - Boehringer Ingelheim Investigational Site, Cainta, Rizal
  - Boehringer Ingelheim Investigational Site, Calamba CIty, Laguna
  - Boehringer Ingelheim Investigational Site, Calamba, Misamis Occidental
  - Boehringer Ingelheim Investigational Site, Calamban City, Laguna
  - Boehringer Ingelheim Investigational Site, Caloocan
  - Boehringer Ingelheim Investigational Site, Camiling, Laguna
  - Boehringer Ingelheim Investigational Site, Cando City, Ilocos Sur
  - Boehringer Ingelheim Investigational Site, Cauayan City, Isabela
  - Boehringer Ingelheim Investigational Site, Cavite City, Cavite
  - Boehringer Ingelheim Investigational Site, Cebu City, Cebu
  - Boehringer Ingelheim Investigational Site, City of Muntinlupa
  - Boehringer Ingelheim Investigational Site, Cruz, Manila
  - Boehringer Ingelheim Investigational Site, Dagupan City, Pangasinan
  - Boehringer Ingelheim Investigational Site, Dasmarinas, Cavite
  - Boehringer Ingelheim Investigational Site, De Vera, Santiago City, Isabela
  - Boehringer Ingelheim Investigational Site, Digolog City, Zamboanga Del Norte
  - Boehringer Ingelheim Investigational Site, Dinalupihan, Bataan
  - Boehringer Ingelheim Investigational Site, Dipolog City, Zamboange Del Norte
  - Boehringer Ingelheim Investigational Site, Ermita, Manila
  - Boehringer Ingelheim Investigational Site, Espana, Manila
  - Boehringer Ingelheim Investigational Site, F Cayco Sampaloc, Manila
  - Boehringer Ingelheim Investigational Site, Gapan City, Nueva Ecija
  - Boehringer Ingelheim Investigational Site, Gingoog City, Misamis Oriental
  - Boehringer Ingelheim Investigational Site, Greenhills, San Juan
  - Boehringer Ingelheim Investigational Site, Guagua, Pampanga
  - Boehringer Ingelheim Investigational Site, Iba, Zambales
  - Boehringer Ingelheim Investigational Site, Ibalong, LegazpiCity, Albay
  - Boehringer Ingelheim Investigational Site, Igano, Molave, Zamboanga Del Sur
  - Boehringer Ingelheim Investigational Site, Ilgan City, Lanao Del Norte
  - Boehringer Ingelheim Investigational Site, Iligan City, Lanao Del Norte
  - Boehringer Ingelheim Investigational Site, Iloilo City, Iloilo
  - Boehringer Ingelheim Investigational Site, Imus, Cavite
  - Boehringer Ingelheim Investigational Site, Kalibo, Aklan
  - Boehringer Ingelheim Investigational Site, Kalookan City, Tala
  - Boehringer Ingelheim Investigational Site, Kaloonkan City
  - Boehringer Ingelheim Investigational Site, Laoag City, Ilocos Norte
  - Boehringer Ingelheim Investigational Site, Laog City, Ilocos Norte
  - Boehringer Ingelheim Investigational Site, Lapu-lapu City, Cebu
  - Boehringer Ingelheim Investigational Site, Las Pina City
  - Boehringer Ingelheim Investigational Site, Las Piñas
  - Boehringer Ingelheim Investigational Site, Legazpi City, Albay
  - Boehringer Ingelheim Investigational Site, Lemery, Batangas
  - Boehringer Ingelheim Investigational Site, Limay, Bataan
  - Boehringer Ingelheim Investigational Site, Lipa City, Batangas
  - Boehringer Ingelheim Investigational Site, Lucena City, Quezon
  - Boehringer Ingelheim Investigational Site, Makati City
  - Boehringer Ingelheim Investigational Site, Malate, Manila
  - Boehringer Ingelheim Investigational Site, Mandaluyong
  - Boehringer Ingelheim Investigational Site, Mandaluyong City, Edsa
  - Boehringer Ingelheim Investigational Site, Marikina City
  - Boehringer Ingelheim Investigational Site, Marilao, Bulacan
  - Boehringer Ingelheim Investigational Site, Masangkay Tondo, Manila
  - Boehringer Ingelheim Investigational Site, Meycauayan, Bulacan
  - Boehringer Ingelheim Investigational Site, Morayta Sampaloc, Manila
  - Boehringer Ingelheim Investigational Site, Munoz City, Nueva Ecija
  - Boehringer Ingelheim Investigational Site, Naga City, Camarines Sur
  - Boehringer Ingelheim Investigational Site, Naga City, Carmarines Sur
  - Boehringer Ingelheim Investigational Site, Olonggapo City, Zambales
  - Boehringer Ingelheim Investigational Site, Ormoc City, Leyte
  - Boehringer Ingelheim Investigational Site, Oroquita City, Misamis Occidental
  - Boehringer Ingelheim Investigational Site, Ozamis City, Misamis Occidental
  - Boehringer Ingelheim Investigational Site, Ozamis City, Misamis
  - Boehringer Ingelheim Investigational Site, Paranaque City
  - Boehringer Ingelheim Investigational Site, Pasay
  - Boehringer Ingelheim Investigational Site, Pasig
  - Boehringer Ingelheim Investigational Site, Pinamalaayan, Calapan City, Oriental Mindoro
  - Boehringer Ingelheim Investigational Site, Pulilan, Bulacan
  - Boehringer Ingelheim Investigational Site, Quezon City
  - Boehringer Ingelheim Investigational Site, Quezon City, Diliman
  - Boehringer Ingelheim Investigational Site, Roxas City, Capiz
  - Boehringer Ingelheim Investigational Site, Roxas, Isabela
  - Boehringer Ingelheim Investigational Site, Sampaloc, Manila
  - Boehringer Ingelheim Investigational Site, San Carlos City, Pangasinan
  - Boehringer Ingelheim Investigational Site, San Fernanado City, Pampanga
  - Boehringer Ingelheim Investigational Site, San Fernando City, La Union
  - Boehringer Ingelheim Investigational Site, San Fernando City, Pampanga
  - Boehringer Ingelheim Investigational Site, San Miguel, Manila
  - Boehringer Ingelheim Investigational Site, San Pablo City, Laguna
  - Boehringer Ingelheim Investigational Site, San Pedro, Laguna
  - Boehringer Ingelheim Investigational Site, Santa Cruz, Laguna
  - Boehringer Ingelheim Investigational Site, Santa Maria, Bulacan
  - Boehringer Ingelheim Investigational Site, Santa Maria, Bulaccan
  - Boehringer Ingelheim Investigational Site, Santiago City, Isabela
  - Boehringer Ingelheim Investigational Site, Sorsogon City, Sorsogon
  - Boehringer Ingelheim Investigational Site, Surigao City, Surigao Del Norte
  - Boehringer Ingelheim Investigational Site, Taal, Batangas
  - Boehringer Ingelheim Investigational Site, Tacloban City, Leyte
  - Boehringer Ingelheim Investigational Site, Taft Ave, Manila
  - Boehringer Ingelheim Investigational Site, Taft, Manila
  - Boehringer Ingelheim Investigational Site, Tagbilaran City, Bohol
  - Boehringer Ingelheim Investigational Site, Tanauan City, Batangas
  - Boehringer Ingelheim Investigational Site, Tarlac City, Tarlac
  - Boehringer Ingelheim Investigational Site, Tondo, Manila
  - Boehringer Ingelheim Investigational Site, Tuguegarao City, Cagayan
  - Boehringer Ingelheim Investigational Site, Urdaneta City, Pangasinan
  - Boehringer Ingelheim Investigational Site, Valenzuela
  - Boehringer Ingelheim Investigational Site, Vigan City, Ilocos Sur
  - Boehringer Ingelheim Investigational Site, Vigan City. Ilocos Sur

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The protocol specified that the study will consist of 16,000 subjects. However, there are only 15, 268 case report forms (CRFs) submitted
Period: Overall Study
Arm/Group | Telmisartan (Micardis)
Started | 15268
Completed | 15113
Not Completed | 155
Not completed — Adverse Event | 5
Not completed — Protocol Violation | 14
Not completed — Lost to Follow-up | 46
Not completed — Other reason not defined above | 90

BASELINE CHARACTERISTICS:
Population: The figure was based on the ITT (intention to treat) population which was reported in the PMS report. The total ITT population is 14, 161.
Arm/Group | Telmisartan (Micardis)
Number analyzed (Participants) | 14161
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age summarized for 13659 subjects and 502 subjects were missing age information
  Years | 59 (9.9)
Gender [Number; unit: Number of participants] — There are 32 subjects with missing gender information
  Number of participants
    Female | 8253
    Male | 5876

OUTCOME MEASURES:

1. Primary Outcome: Response Rate at the End of 30 Day Period
Description: Response rate of Blood Pressure assessed in the following categories:
  * Sitting SBP < 130 mmHg and/or a reduction of > 20 mmHg from baseline
  * Sitting DBP < 85 mmHg and/or a reduction of > 10 mmHg from baseline Sitting BP normalization < 130 mmHg and DBP < 85 mmHg
Time Frame: End of 30 day Period
Population: ITT Population: all patients who took at least one dose of the study medication and have at least one point treatment efficacy data available
Measure: Number; unit: Percentage of patients
Arm/Group | Telmisartan (Micardis)
Number analyzed (Participants) | 14161
Percentage of patients
  Sitting SBP response | 41.4
  Sitting DBP response | 66.3
  Sitting BP normalization | 31.2

2. Primary Outcome: Response Rate at the End of 60 Day Period
Description: Response rate on Blood Pressure:
  1. Sitting SBP < 130 mmHg and/or a reduction of > 20 mmHg from baseline.
  2. Sitting DBP < 85 mmHg and/or a reduction of > 10 mmHg from baseline.
  3. Sitting BP normalization < 130 mmHg and DBP < 85 mmHg
Time Frame: At the end of 60 day period
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Telmisartan (Micardis)
Number analyzed (Participants) | 14161
Percentage of patients
  Sitting SBP response | 75.5
  Sitting DBP response | 88.1
  Sitting BP normalization | 69.1

3. Primary Outcome: Change in Systolic Blood Pressure (SBP) From Baseline
Description: Change in SBP = Value in visit 1(baseline) minus value in visit 3 (at 60-day treatment period)
Time Frame: Baseline and 60 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Telmisartan (Micardis)
Number analyzed (Participants) | 14161
mmHg | 30.2 (15.4)

4. Primary Outcome: Change in Diastolic Blood Pressure (DBP) From Baseline
Description: Change in DBP = Value in visit 1(baseline) minus value in visit 3 (at 60-day treatment period)
Time Frame: Baseline and 60 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Telmisartan (Micardis)
Number analyzed (Participants) | 14161
mmHg | 15.9 (10)

5. Secondary Outcome: Percentage of Patients With Presence of Metabolic Risk Factor
Description: Presence of metabolic risk factor was identified by the existence of 3 out of the 5 risk factors namely:
  a.) presence of diabetes mellitus; b) presence of dyslipidemia; c) presence of albuminuria; d) presence of ventricular hypertrophy; and e) presence of co-morbidities,
  based on patients' Medical History
Time Frame: At the end of 60 day period
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Telmisartan (Micardis)
Number analyzed (Participants) | 14161
Percentage of patients | 20.0

ADVERSE EVENTS:
Time Frame: Upto 60 Days
Arm/Group | Telmisartan (Micardis)
Serious Adverse Events (participants affected / at risk) | 5/15268
Other Adverse Events (participants affected / at risk) | 0/15268
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telmisartan (Micardis) (N=15268)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 2
DIARRHEA (Gastrointestinal disorders) | 1
HIGH BLOOD PRESSURE (190/120) (Investigations) | 1
MASSIVE HEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.